CLINICAL TRIAL: NCT06358716
Title: Glycaemic Index Determination in Oral Nutrition Supplements
Acronym: BEGINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de Lleida (Other)
Collaborators: Lactalis (Industry)
Responsible Party: Principal Investigator, José Serrano, Professor, Universitat de Lleida
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CEIC-3037
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Glucose Metabolism Disorders
Keywords: Glycemic index; Glucose; Post-prandial; Digestible carbohydrates
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Oral Nutritional Supplement 1 (Experimental): Oral Nutritional Supplement 1
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 1
- Oral Nutritional Supplement 2 (Experimental): Oral Nutritional Supplement 2
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 2
- Oral Nutritional Supplement 3 (Experimental): Oral Nutritional Supplement 3
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 3
- Oral Nutritional Supplement 4 (Experimental): Oral Nutritional Supplement 4
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 4
- Oral Nutritional Supplement 5 (Experimental): Oral Nutritional Supplement 5
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 5
- Oral Nutritional Supplement 6 (Experimental): Oral Nutritional Supplement 6
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 6
- Oral Nutritional Supplement 7 (Experimental): Oral Nutritional Supplement 7
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 7
- Oral Nutritional Supplement 8 (Experimental): Oral Nutritional Supplement 8
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 8
- Oral Nutritional Supplement 9 (Experimental): Oral Nutritional Supplement 9
  Interventions: Dietary Supplement: Complete Oral Nutrition Supplement 9
- Glucose (Active Comparator): Glucose solution
  Interventions: Dietary Supplement: Glucose

INTERVENTIONS:
Dietary Supplement: Complete Oral Nutrition Supplement 1 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 1
Dietary Supplement: Complete Oral Nutrition Supplement 2 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 2
Dietary Supplement: Complete Oral Nutrition Supplement 3 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 3
Dietary Supplement: Complete Oral Nutrition Supplement 4 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 4
Dietary Supplement: Complete Oral Nutrition Supplement 5 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 5
Dietary Supplement: Complete Oral Nutrition Supplement 6 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 6
Dietary Supplement: Complete Oral Nutrition Supplement 7 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 7
Dietary Supplement: Complete Oral Nutrition Supplement 8 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 8
Dietary Supplement: Complete Oral Nutrition Supplement 9 — Liquid formula produced by several food ingredients to provide a balance nutrient intake
  Arms: Oral Nutritional Supplement 9
Dietary Supplement: Glucose — 25 mg of glucose dissolved in 200 mL
  Arms: Glucose

SUMMARY:
The glycemic index is the ability of carbohydrates in foods to induce increases in blood glucose levels after consuming them. Based on the capacity for increasing blood glucose levels, foods can be classified as having a low, medium, or high glycemic index. This property is of interest in health and nutrition because it allows estimating the impact the food will have on postprandial glycemia, which may able better food selection in situations where adequate glycemic control is required, such as in individuals diagnosed with Diabetes Mellitus. The objective of this study is to determine the glycemic index of 9 formulations of complete oral nutrition supplements and classify them based on their glycemic response.

DETAILED DESCRIPTION:
The determination of the glycemic index will be conducted following the protocol described in the International Standard Organization 26642. Specifically, the glycemic response of each food will be determined in 15 healthy volunteers, using a glucose-containing beverage with 25 g of glucose in 200 mL as a control for glycemic response measurement. The amount of food each volunteer will test will be equivalent to an intake of 25 g of digestible carbohydrates in a single intake. Subsequently, increases in blood glucose levels will be recorded at 15, 30, 45, 60, 90, and 120 minutes after initiating the food intake. Blood glucose measurements will be performed using a portable glucometer via capillary blood. The area under the curve of the increase in glucemia will be estimated using the trapezoidal method, and these will be compared with the glucose increases provided by the glucose-containing beverage.

ELIGIBILITY:
Inclusion Criteria:

• Healthy volunteers with no known food allergy or intolerance and pharmacological treatments known to affect glucose tolerance (excluding oral contraceptives)

Exclusion Criteria:

* Known history of diabetes mellitus or the use of antihyperglycemic drugs or insulin to treat diabetes and related conditions.
* Any acute, chronic disease or any other serious complications that may interfere with glucose metabolism.
* Subjects using any medication (eg steroids, protease inhibitors or antipsychotics, etc.) that would interfere with the digestion and nutrient absorption.
* Subjects having gastrointestinal diseases that may interfere with nutrient absorption, distribution, metabolism, excretion
* A major medical or surgical event requiring hospitalization within the preceding 3 months.
* Pregnancy

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index | Post-prandial until 120 minutes after food intake
  The area under the curve of glucose levels after the post-prandial intake of the oral nutrition supplement compared with the area under the curve of glucose levels after a post-prandial intake of a glucose solution

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lleida, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No